CLINICAL TRIAL: NCT03908892
Title: A Clinical Study on the Treatment of Paronychia Caused by Afatinib With Zanthoxylum Nitidum Tincture
Brief Title: Effect of Zanthoxylum Nitidum Tincture for Paronychia Caused by Afatinib
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangzhou University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Haibo Zhang, Professor, Guangzhou University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019KT1122
Record Dates: First submitted 2019-02-21; First posted 2019-04-09 (Actual); Last update posted 2022-08-15 (Actual); Status verified 2022-08

CONDITIONS: Paronychia
Keywords: Paronychia; Zanthoxylum nitidum tincture; Afatinib
MeSH Terms: conditions — Paronychia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combination group (Experimental): Local use of 1% tetracycline ointment for the sick nail(s), 3 times a day, plus local application with zanthoxylum nitidum tincture soaked blocks for the sick nail(s) for 30 minutes, twice a day, till paronychia relief or progression.
  Interventions: Drug: zanthoxylum nitidum tincture; Drug: tetracycline ointment
- Control group (Active Comparator): Local use of 1% tetracycline ointment for the sick nail(s), 3 times a day, till paronychia relief or progression.
  Interventions: Drug: tetracycline ointment

INTERVENTIONS:
Drug: zanthoxylum nitidum tincture — Local application with zanthoxylum nitidum tincture soaked blocks for the sick nail(s) for 30 minutes, twice a day.
  Arms: Combination group
Drug: tetracycline ointment — Local use of 1% tetracycline ointment for the sick nail(s), 3 times a day

SUMMARY:
This is a randomized control trial evaluating the efficacy of zanthoxylum nitidum tincture on preventing progression of paronychia caused by afatinib from grade 1 to grade 2/3. Enrolled participates will randomly receive original treatment or original treatment plus zanthoxylum nitidum tincture immersion of the sick nail(s).

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically or cytologically confirmed non-small cell lung cancer；
2. Undergoing treatment with afatinib；
3. With grade 1 paronychia；
4. Age between 18 to 80 years old；
5. Estimated life expectancy of more than months；
6. With the written informed consent.

Exclusion Criteria:

1. Paronychia before afatinib treatment;
2. Grade 2 or severer paronychia;
3. Stop using afatinib or with reduced dose of afatinib;
4. Currently diagnosed with severe encephalopathy or psychiatric disorders affecting patients ability of self expression.
5. Has other legal, medical or ethical reasons that patients are not appropriate for clinical study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2019-06-12 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Paronychia progress rate | Through study completion, an average of 10 days.
  Incidence of grade 2 or more paronychia during paronychia treatment period will be reported. This period will be from randomization till paronychia relief or progression. Frequency of evaluation for paronychia will be everyday.

SECONDARY OUTCOMES:
Time to paronychia progress | Through study completion, an average of 10 days.
  The time elapsed from randomization to either the date of grade 2 or more paronychia occurrence, treatment completion, or last follow-up information. Frequency of evaluation for paronychia will be everyday.
Time to paronychia relief | Through study completion, an average of 10 days.
  The time elapsed from randomization to either the date of paronychia relief, treatment completion, or last follow-up information. Paronychia relief is defined as that paronychia disappears. Frequency of evaluation for paronychia will be everyday.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Provincial Hospital of Chinese Medicine, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No